CLINICAL TRIAL: NCT02491268
Title: A Trial of Cilostazol for Prevention of Conversion From Mild Cognitive Impairment to Dementia
Brief Title: A Trial of Cilostazol in Patients With Mild Cognitive Impairment (COMCID)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cerebral and Cardiovascular Center, Japan (Other)
Responsible Party: Principal Investigator, Masafumi Ihara, Chief Physician (Head of Neurology), National Cerebral and Cardiovascular Center, Japan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TRINEU1321
Record Dates: First submitted 2015-07-01; First posted 2015-07-08 (Estimated); Last update posted 2020-12-04 (Actual); Status verified 2020-12

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Cilostazol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cilostazol 50mg B.I.D. (Experimental): After the registration, the Site Investigators should start protocol treatment within 28 days including the day of registration.
  Protocol treatment defines as follows;
  Investigational Treatment:
  Cilostazol 50mg B.I.D. p.o. 96 Weeks
  Interventions: Drug: Cilostazol
- Placebo B.I.D. (Placebo Comparator): After the registration, the Site Investigators should start protocol treatment within 28 days including the day of registration.
  Protocol treatment defines as follows;
  Comparative Treatment:
  Placebo B.I.D. p.o. 96 Weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cilostazol
  Arms: Cilostazol 50mg B.I.D.
Drug: Placebo
  Arms: Placebo B.I.D.

SUMMARY:
Epidemiological, clinicopathological and animal studies show that vascular disease in various forms contributes to cognitive decline. Increasing age is the strongest risk for dementia irrespective of whether it results from a vascular etiology or neurodegenerative disease processes such as in Alzheimer's disease (AD). AD and vascular cognitive impairment, the two most common causes of dementia, represent two extremes of a spectrum of disorders; however, a number of entities, which possess varying degrees of neurodegenerative and vascular pathologies, occur in between. The pure forms of the disorders are preferred for convenience to label, treat or manage but conditions within the spectrum are the norm rather than the exception as dementia advances. Therefore, combinatorial therapy directed at both vascular and neurodegenerative aspects of dementia is a promising approach for the treatment of dementia in the elderly.

Cilostazol acts as an antiplatelet agent and has other pleiotropic effects based on phosphodiesterase-3-dependent mechanisms. Increasing evidence suggests that cilostazol offers endothelial protection, via pleiotropic effects. Intriguingly, cilostazol has been shown to decrease amyloid beta (Abeta) accumulation and protect Abeta-induced cognitive deficits in an experimental model. In a pilot study of 10 patients with moderate AD (mean MMSE score, 11.9 points) who received donepezil, cilostazol add-on treatment for 5-6 months demonstrated significantly increased MMSE score in comparison to baseline. Moreover, cilostazol was shown to be effective in preventing cognitive decline in patients with AD with cerebrovascular diseases, mild cognitive impairment (MCI), and mild dementia who received donepezil.

These results highlight the need for a comprehensive prospective cohort study to analyze the effect of cilostazol on the preservation of cognitive function in patients with early-stage cognitive impairment, namely MCI.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 55-84 (inclusive)
2. Study partner who sufficiently knows the daily life of the patient
3. Patients with MCI who satisfy the core clinical criteria of National Institute for Aging-Alzheimer Association for MCI (nearly equivalent to mild neurocognitive disorder in Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition) and who also satisfy the following three criteria:

   i) Memory complaint by subject or study partner Type I: Memory complaint by subject that is verified by a study partner Type II: Otherwise, memory complaint by study partner with the evidence of memory impairment Note) Memory complaint by subject that is not verified by study partner will be excluded.

   ii) Mini-Mental State Examination (MMSE) scores between 22 and 28 (inclusive) iii) Clinical Dementia Rating (CDR) = 0.5
4. Written informed consent provided for study participation

Exclusion Criteria:

1. Parkinson's disease, Huntington's disease, normal pressure hydrocephalus, progressive supranuclear palsy, epilepsy, multiple sclerosis, cerebral infection, or subsequent complication caused by head trauma.
2. Findings of multiple infarction, brain tumor, or subdural hematoma on MRI performed within 48 weeks before provisional registration.
3. Contraindications for MRI such as magnetic body or metal.
4. History of major depression or bipolar disorder within 48 weeks before provisional registration, alcohol or other substance abuse within 96 weeks before provisional registration, other diseases or unstable conditions.
5. Poorly controlled diabetes mellitus (HbA1c>9.0%).
6. Cognitive impairment due to deficiency of vitamin B12 or folate.
7. Neurosyphilis.
8. Cognitive impairment due to thyroid function abnormality.
9. Psychoactive drugs within 4 weeks before provisional registration.
10. Oral anticoagulants within 4 weeks before provisional registration.
11. Double antiplatelet therapy (cf. Aspirin, Clopidogrel but not Cilostazol) within 4 weeks before provisional registration.
12. Poorly controlled diabetes mellitus treated with insulin within 4 weeks before provisional registration.
13. Episode of hypoglycemic attack with loss of consciousness within 4 weeks before provisional registration.
14. Anti-dementia drugs within 4 weeks before provisional registration.
15. Participation in any other new drug study for Alzheimer's disease.
16. Current bleeding or bleeding disorders.
17. Congestive heart failure.
18. Coronary artery stenosis.
19. Sustained high blood pressure within 2 weeks before provisional registration.
20. History of drug hypersensitivity to Cilostazol.
21. The subject or the subject's spouse pregnant or breast-feeding at the time of provisional registration.
22. Difficulty in neuropsychological tests due to hearing or visual impairment.
23. Considered by the principal investigator to be ineligible.

Ages: 55 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2020-08-14 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Mini Mental State Examination (MMSE) | 96 weeks

SECONDARY OUTCOMES:
Conversion from MCI to All-cause Dementia | up to 96 weeks
  Dementia is diagnosed clinically when the patient meets core clinical criteria for dementia with reference to Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition.
Cognitive Decline on Clinical dementia rating-sum of boxes (CDR-SB) | baseline, 48 weeks, and 96 weeks
Cognitive Decline on Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-Cog) 14 | baseline, 48 weeks, and 96 weeks
Cognitive Decline on Logical Memory subtest of the Wechsler Memory Scale-Revised (WMS-R) | baseline, 48 weeks, and 96 weeks
Functional Decline on Alzheimer's disease Cooperative Study scale for activities of daily living in MCI (ADCS-MCI-ADL) | baseline, 48 weeks, and 96 weeks
Hippocampal volume | baseline and 96 weeks
  Magnetization prepared rapid acquisition with gradient echo is used to assess hippocampal volume.

OTHER OUTCOMES:
Cognitive Decline on Free and Cued Selective Reminding Test (FCSRT) | baseline, 48 weeks, and 96 weeks
Cognitive Decline on Trail making test (TMT) | baseline, 48 weeks, and 96 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- National Cerebral and Cardiovascular Center, Suita, Osaka, Japan

REFERENCES:
- [Derived] Saito S, Suzuki K, Ohtani R, Maki T, Kowa H, Tachibana H, Washida K, Kawabata N, Mizuno T, Kanki R, Sudoh S, Kitaguchi H, Shindo K, Shindo A, Oka N, Yamamoto K, Yasuno F, Kakuta C, Kakuta R, Yamamoto Y, Hattori Y, Takahashi Y, Nakaoku Y, Tonomura S, Oishi N, Aso T, Taguchi A, Kagimura T, Kojima S, Taketsuna M, Tomimoto H, Takahashi R, Fukuyama H, Nagatsuka K, Yamamoto H, Fukushima M, Ihara M; COMCID Trial Investigator Group. Efficacy and Safety of Cilostazol in Mild Cognitive Impairment: A Randomized Clinical Trial. JAMA Netw Open. 2023 Dec 1;6(12):e2344938. doi: 10.1001/jamanetworkopen.2023.44938. PMID 38048134